CLINICAL TRIAL: NCT06777095
Title: Effects of Different Kinesio Taping Treatments Added to the Physical Therapy Program on Pain, Endurance, Lumbar Proprioception, Mobility and Disability in Patients Diagnosed With Lumbar Disc Herniation: A Randomized Controlled Trial
Brief Title: Effects of Kinesio Taping on Pain, Endurance, Proprioception, Mobility and Disability in Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sevtap Günay (Other)
Responsible Party: Sponsor-Investigator, Sevtap Günay, Associate Professor, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Izmir Katip Celebi
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Disc Herniation; Lumbar Disc Disease; Chronic Pain
Keywords: Taping; Low back pain; Lumbar disc herniation; Muscular fitness; Proprioception; Mobility; Disability
MeSH Terms: conditions — Intervertebral Disc Displacement; Intervertebral disc disease; Chronic Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients participating in the study were not informed about taping methods. The assessor was blinded as there was no taping and the assessor did not know which group the participant was in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): In addition to routine physical therapy sessions, I taping was applied to the paraspinal muscles.
  Interventions: Other: Routine Treatment + I Taping
- Group 2 (Active Comparator): In addition to routine physical therapy sessions, star taping was applied to sensitive points.
  Interventions: Other: Routine Treatment + Star Taping
- Group 3 (Other): No application (no taping) was made outside of the routine physical therapy program.
  Interventions: Other: Routine Treatment

INTERVENTIONS:
Other: Routine Treatment + I Taping — Routine physical therapy program (10 sessions of hotpack, Transcutaneous electrical nerve stimulation (TENS), and ultrasound every day for 2 weeks) was applied. In addition to routine treatment, I taping (a total of 5 times every 3 days) was performed. Two I-shaped kinesio tapings were applied on the paraspinal muscles from the posterior superior iliac spine to the T12 level. 50% tension was applied to the area of the tapes outside the anchor points.
  Arms: Group 1
Other: Routine Treatment + Star Taping — Routine physical therapy program (10 sessions of hotpack, Transcutaneous electrical nerve stimulation (TENS), and ultrasound every day for 2 weeks) was applied. In addition to routine treatment, star taping (a total of 5 times every 3 days) was performed. Four I tapes, one vertical, one horizontal and two at a 45° angle to the vertical tape, were applied to the point of maximum pain in the lumbar region. 25% tension was applied to the midpoint of the tapes except for the ends.
  Arms: Group 2
Other: Routine Treatment — Routine physical therapy program (10 sessions of hotpack, Transcutaneous electrical nerve stimulation (TENS), and ultrasound every day for 2 weeks) was applied. No taping was applied.
  Arms: Group 3

SUMMARY:
In addition to the physical therapy program, taping was applied to 90 patients diagnosed with lumbar disc herniation. 90 patients were randomized into 3 groups. Group 1 received star-shaped taping to the lumbar region in addition to physical therapy, Group 2 received I-shaped taping to the erector spinae muscles in addition to physical therapy, and Group 3 was planned as the control group. In the first evaluation, sociodemographic information and disease duration (months) were questioned. Then, pain, muscle strength and endurance mobility, lumbar proprioception, functional level, and disability were evaluated. Evaluations were performed before treatment, after taping and at the end of the 12th week.

DETAILED DESCRIPTION:
The study included 90 patients aged between 18-65 years who were diagnosed with LDH by magnetic resonance imaging (MRI), had moderate to severe low back pain (Numeric Rating Scale >4) for at least 6 weeks, and were planned to receive a physical therapy program (10 sessions of hotpack, Transcutaneous electrical nerve stimulation (TENS), and ultrasound every day for 2 weeks). The 90 patients included in the study were randomized into 3 groups using the computer-assisted randomization method. Group 1 received star-shaped taping to the lumbar region in addition to physical therapy (5 times in total every 3 days), Group 2 received I-shaped taping to the erector spinae muscles in addition to physical therapy (5 times in total every 3 days), and Group 3 was planned as the control group. In the first evaluation, sociodemographic information (age, gender, height (m), weight (kg), BMI (kg/m2)) and disease duration (months) were questioned. Then, pain (pain intensity and pressure pain threshold), muscle strength (lumbar extensor muscle strength) and endurance (trunk extensor muscle endurance), mobility (lumbar lordosis angle, joint range of motion), lumbar proprioception, functional level, disability evaluations were performed. Evaluations were performed before treatment, after the taping application and at the end of the 12th week. Post-treatment evaluations were performed the day after the tape was removed.

ELIGIBILITY:
Inclusion Criteria:

* Having moderate to severe low back pain (Numeric Rating Scale>3) for at least 6 weeks
* Voluntariness to participate in the study

Exclusion Criteria:

* History of lumbar fracture or tumor
* Previous lumbosacral or abdominal surgery
* Ankylosing spondylitis, spondylolisthesis, fibromyalgia, peripheral neurogenic disease
* Pregnancy
* History of cancer
* Demonstrated allergy/intolerance to kinesiotaping during a test performed before the initial evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Pain intensity assessment | Baseline, day after last taping application (week 2), 12 weeks after baseline
  Pain intensity was measured using the Pain Intensity Numerical Rating Scale, which is most commonly used in the management of patients with chronic low back pain. The scale has 11 points ranging from no pain = 0 to worst possible pain = 10. Patients were asked to indicate their pain intensity during the "last 24 hours" or "average pain" at rest.
Pressure pain threshold assessment | Baseline, day after last taping application (week 2), 12 weeks after baseline
  The pressure pain threshold was determined in kg/cm2 using an algometer device. Measurements were made at 4 points, 5 cm lateral to the L3 and L5 spinous processes on the right and left. The patient was informed to give the command 'stop' when the pressure sensitivity became unbearable or turned into pain. The test was stopped as soon as the patient reported pain and the applied force was recorded. 2 measurements were made at 30-second intervals and the average of the measurements was used. If the participant did not report pain at a force equivalent to 100 N/s, the test was stopped and this value was accepted.
Muscle strength assessment | Baseline, day after last taping application (week 2), 12 weeks after baseline
  Lumbar extensor muscle strength was measured with a hand held dynamometer. Participants were positioned face down on a stretcher with their hands clasped. The base of the dynamometer was fixed to the center of the T4 spine and participants were asked to extend their trunks. The tests were repeated twice with at least a one-minute rest. The higher value was recorded as the result.
Endurance assessment | Baseline, day after last taping application (week 2), 12 weeks after baseline
  The measurement was made using the Biering-Sorensen test. The participant placed the upper half of his/her body on another examination table at a lower height. The participant was asked to hold his/her body isometrically in a horizontal position with hands clasped behind the head until fatigue or pain was felt. The test was terminated when any part of the participant's upper extremities touched the table. The tests were repeated twice with at least a one-minute rest break. The higher value was recorded as the result.
Lumbar lordosis angle assessment | Baseline, day after last taping application (week 2), 12 weeks after baseline
  Lumbar lordosis was measured using a digital inclinometer. The participant stood with their feet 15 cm apart and their arms at their sides while looking ahead. In this position, the T12-L1 and S1 spine levels were marked by the physiotherapist. Lumbar lordosis was calculated by placing one end of the inclinometer on T12-L1 and the other on the sacrum.
Lumbar joint range of motion assessment | Baseline, day after last taping application (week 2), 12 weeks after baseline
  Participants' lumbar flexion, extension and lateral flexion active joint range of motion measurements were evaluated angularly with a universal goniometer.
Proprioception assessment | Baseline, day after last taping application (week 2), 12 weeks after baseline
  Proprioception was assessed by having the participants attempt to reproduce the target position. Three different target positions were selected. The participants were asked to repeat two different trunk positions from upright posture to 45° and 60° flexion with the eyes looking forward, and one position to 15° extension. Each participant was positioned in 45° lumbar flexion for 10 seconds after a neutral starting position and was asked to remember this position. The participant then returned to the neutral position and was given verbal instructions to reproduce the target position as accurately as possible. The participant reported to the therapist that he had reached the target position as perceived. The participant was asked to maintain the final position for 3 seconds and this position was recorded. The same procedures were repeated for 60° lumbar flexion and 15° lumbar extension. Each trial was repeated three times with a 30-second rest; the mean was then calculated.
Functional level assessment | Baseline, day after last taping application (week 2), 12 weeks after baseline
  A 30-second stand-up-sit test was performed to determine the functional level. Participants were asked to sit in a back-supported chair without arm support, with their hands crossed on their shoulders. Participants were asked to sit immediately after coming to an upright standing position. A trial test was performed to learn the test. The individual who learned the test was asked to sit down and stand up for 30 seconds and the number of repetitions of the movement was recorded.
Disability assessment | Baseline, day after last taping application (week 2), 12 weeks after baseline
  The Roland Morris Disability Questionnaire was used to assess disability due to low back pain. The questionnaire consists of 24 items regarding physical activity, rest/sleep, psychosocial outcomes, home management, nutrition, and pain frequency. Higher scores indicate increasing disability.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Meryem SERTPOYRAZ, Assoc. Dr., Study Director — Department of Physiotherapy and Rehabilitation, Bakircay University Training and Research Hospital; Hilal UZUNLAR, PhD(c), RA, Study Chair — Izmir Katip Çelebi University, Department of Physiotherapy and Rehabilitation; Ecem SAK, Ass.Dr., Study Chair — Department of Physiotherapy and Rehabilitation, Bakircay University Training and Research Hospital
Locations (1):
- Izmir Bakircay University Cigli Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreiner DS, Hwang SW, Easa JE, Resnick DK, Baisden JL, Bess S, Cho CH, DePalma MJ, Dougherty P 2nd, Fernand R, Ghiselli G, Hanna AS, Lamer T, Lisi AJ, Mazanec DJ, Meagher RJ, Nucci RC, Patel RD, Sembrano JN, Sharma AK, Summers JT, Taleghani CK, Tontz WL Jr, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of lumbar disc herniation with radiculopathy. Spine J. 2014 Jan;14(1):180-91. doi: 10.1016/j.spinee.2013.08.003. Epub 2013 Nov 14. PMID 24239490
- [Background] Keles BY, Yalcinkaya EY, Gunduz B, Bardak AN, Erhan B. Kinesio Taping in patients with lumbar disc herniation: A randomised, controlled, double-blind study. J Back Musculoskelet Rehabil. 2017;30(3):543-550. doi: 10.3233/BMR-150491. PMID 27858685
- [Background] Hayden JA, van Tulder MW, Malmivaara A, Koes BW. Exercise therapy for treatment of non-specific low back pain. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD000335. doi: 10.1002/14651858.CD000335.pub2. PMID 16034851
- [Background] Suzuki H, Aono S, Inoue S, Imajo Y, Nishida N, Funaba M, Harada H, Mori A, Matsumoto M, Higuchi F, Nakagawa S, Tahara S, Ikeda S, Izumi H, Taguchi T, Ushida T, Sakai T. Clinically significant changes in pain along the Pain Intensity Numerical Rating Scale in patients with chronic low back pain. PLoS One. 2020 Mar 3;15(3):e0229228. doi: 10.1371/journal.pone.0229228. eCollection 2020. PMID 32126108
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] de Oliveira RF, Liebano RE, Costa Lda C, Rissato LL, Costa LO. Immediate effects of region-specific and non-region-specific spinal manipulative therapy in patients with chronic low back pain: a randomized controlled trial. Phys Ther. 2013 Jun;93(6):748-56. doi: 10.2522/ptj.20120256. Epub 2013 Feb 21. PMID 23431209
- [Background] Karthikbabu S, Chakrapani M. Hand-Held Dynamometer is a Reliable Tool to Measure Trunk Muscle Strength in Chronic Stroke. J Clin Diagn Res. 2017 Sep;11(9):YC09-YC12. doi: 10.7860/JCDR/2017/28105.10672. Epub 2017 Sep 1. PMID 29207821
- [Background] Latimer J, Maher CG, Refshauge K, Colaco I. The reliability and validity of the Biering-Sorensen test in asymptomatic subjects and subjects reporting current or previous nonspecific low back pain. Spine (Phila Pa 1976). 1999 Oct 15;24(20):2085-9; discussion 2090. doi: 10.1097/00007632-199910150-00004. PMID 10543003
- [Background] Chang NJ, Chou W, Hsiao PC, Chang WD, Lo YM. Acute effects of Kinesio taping on pain, disability and back extensor muscle endurance in patients with low back pain caused by magnetic resonance imaging-confirmed lumbar disc degeneration. J Back Musculoskelet Rehabil. 2018 Feb 6;31(1):85-93. doi: 10.3233/BMR-169681. PMID 28800306
- [Background] Abbasi S, Hadian Rasanani MR, Ghotbi N, Olyaei GR, Bozorgmehr A, Rasouli O. Short-term effect of kinesiology taping on pain, functional disability and lumbar proprioception in individuals with nonspecific chronic low back pain: a double-blinded, randomized trial. Chiropr Man Therap. 2020 Nov 20;28(1):63. doi: 10.1186/s12998-020-00349-y. PMID 33213492
- [Background] Lin YH, Sun MH. The effect of lifting and lowering an external load on repositioning error of trunk flexion-extension in subjects with and without low back pain. Clin Rehabil. 2006 Jul;20(7):603-8. doi: 10.1191/0269215506cr971oa. PMID 16894803
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Kucukdeveci AA, Tennant A, Elhan AH, Niyazoglu H. Validation of the Turkish version of the Roland-Morris Disability Questionnaire for use in low back pain. Spine (Phila Pa 1976). 2001 Dec 15;26(24):2738-43. doi: 10.1097/00007632-200112150-00024. PMID 11740366
- [Background] Alahmari KA, Rengaramanujam K, Reddy RS, Samuel PS, Tedla JS, Kakaraparthi VN, Ahmad I. The immediate and short-term effects of dynamic taping on pain, endurance, disability, mobility and kinesiophobia in individuals with chronic non-specific low back pain: A randomized controlled trial. PLoS One. 2020 Sep 29;15(9):e0239505. doi: 10.1371/journal.pone.0239505. eCollection 2020. PMID 32991582
- [Derived] Altas EU, Uzunlar H, Beytorun E, Danaci EC, Sertpoyraz FM, Ucurum SG. Effects of different kinesiology taping applications on Pain, muscular Fitness, Proprioception, Mobility, Functionality, and disability in patients with lumbar disc herniation. Ir J Med Sci. 2026 Jan 9. doi: 10.1007/s11845-025-04250-6. Online ahead of print. PMID 41511609